CLINICAL TRIAL: NCT03356353
Title: Sildenafil for the Prevention of Right Heart Failure Following Continuous-Flow Left Ventricular Assist Device Implantation (The REVAD Study)
Brief Title: Sildenafil for the Prevention of Right Heart Failure Following LVAD Implantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RVD102017
Record Dates: First submitted 2017-11-22; First posted 2017-11-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: End Stage Heart Failure
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: This is an open label single arm trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sildenafil citrate (Experimental): Following enrolment, participants will be given an initial dose of sildenafil 20 mg. If tolerated, a schedule of 20 mg three times daily (tid) will be initiated. Dosage will be titrated over 3-4 days to the target dose of 40 mg tid. If the initial dose is not tolerated, the participant will be exited from the trial.
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate — 20 mg tablets
  Other Names: Revatio

SUMMARY:
Continuous-flow left ventricular assist devices (LVAD) move blood from the left ventricle (the largest chamber of the heart) to the aorta (the body's main artery) to help the heart better meet the needs of the body and to improve survival for patients with advanced heart failure (HF). The ability of the right ventricle (the large chamber on the right side of the heart) to keep up with the improved blood flow following LVAD greatly effects how well a person does following surgery. It is understood that a high pulmonary artery pressure (pressure in the blood vessel that takes blood from the right side of the heart to the lungs) measured before surgery, indicates that a higher risk of right heart failure exists after LVAD implantation.

This is important because right heart failure after surgery is related to longer intensive care unit (ICU) and hospital stays, increased morbidity (other health problems) including organ failure and worse outcomes following heart transplant, and increased death rates.

Sildenafil (Revatio®) has been approved by Health Canada in the treatment of pulmonary arterial hypertension (high blood pressure in the lungs) in patients with connective tissue disease. Sildenafil has not yet been approved by Health Canada for the treatment of pulmonary hypertension in heart failure. Sildenafil lowers blood pressure in the lungs and lessens the workload of the right ventricle (the right side of the heart). The purpose of this study is to determine if lowering blood pressure in the lungs, in heart failure patients at risk for developing right heart failure after LVAD implant, lowers the incidence of right heart failure, shortens ICU and hospital stays and reduces morbidity (other health problems) and mortality (death rates).

This is an open label, single arm study. Everyone who participates in this study will receive sildenafil before and after LVAD surgery. It is expected that 24 patients who are scheduled to have LVAD implantation for advanced heart failure will be enrolled from 6 sites across Canada. Participants will be followed in the study for about 2 months.

DETAILED DESCRIPTION:
Initially implanted as a bridge to transplantation, LVADs are increasingly used for the purpose of destination therapy. About 250 patients/year will receive LVAD device therapy in 12 implanting Canadian centres. Outcomes after LVAD implantation are critically dependent on right ventricular (RV) function. Development of right heart failure (RHF) in LVAD patients has a direct effect on mortality and is associated with a prolonged length of intensive care unit (ICU) and hospital admission. RHF in LVAD patients leads to increased morbidity and is associated with worse outcomes after cardiac transplantation. Despite improvements in surgical and medical management the incidence of RHF after LVAD implantation has plateaued at approximately 20-30%. A critical concept in the prevention of post-operative complications involves appropriate patient selection and prophylactic measures directed toward risk factors for development of RHF. To mitigate the risk of RHF after LVAD implantation, many implanting centres are increasingly utilizing pulmonary vasodilating agents in the post-operative period. Despite little evidence to support this approach, the phosphodiesterase-5A (PDE5) inhibitor Sildenafil is now empirically administered for reduction of PVR in some centres after LVAD implantation. Duration of therapy varies but may extend beyond 3 months and in some cases may continue indefinitely or until the time of heart transplant. A small, single-centre, open label study demonstrated that Sildenafil effectively reduced PVR in LVAD patients with persistent pulmonary hypertension post-operatively, however only hemodynamic endpoints were examined. Importantly, the investigation of this strategy was limited to those with elevated PAP, irrespective of their clinical condition or pre-implantation hemodynamic profile. There is a clear need for further research to establish the safety and efficacy of pulmonary vasodilators to either treat or prevent RHF in the LVAD patient population.

The investigators hypothesize that the vasodilatory effects of sildenafil can prevent or reverse the effects of elevated RV afterload and consequent RHF following LVAD implantation, and that preoperative initiation of therapy in an at-risk population is feasible and will be well tolerated. As such, there is a large potential for sildenafil to meet an unmet therapeutic need for patients following LVAD implantation.

The primary objective of this pilot study is to evaluate the tolerability and efficacy of sildenafil therapy initiated prior to and continued after LVAD implantation for the purpose of reducing PVR in patients at increased risk for development of RHF by INTERMACS criteria. The feasibility of introducing sildenafil in this clinical setting along with the ability to reduce PVR will be assessed.

Secondary Objectives: a) To determine the efficacy of sildenafil to reduce the need for prolonged inotropic support and post-operative ICU admission duration b) To determine the tolerability and feasibility of the proposed dosing strategy c) To determine the impact of sildenafil therapy on renal function and systemic arterial blood pressure d) To assess the impact of sildenafil therapy on the likelihood of development of post-operative RHF by INTERMACS criteria

STUDY METHODS:

1. Single-arm, open-label, prospective, multi-centre, interventional, feasibility and efficacy, pilot study of sildenafil in patients undergoing LVAD implantation.
2. This multi (6)-centre, Canadian trial is investigator initiated and industry sponsored. The study design, coordination and conduction and other study tasks including monitoring will be performed by the study investigators.

Following enrolment into the study, subjects will have their data (i.e. weight, blood pressure, pulse, lab work, medications, RHC data, ECG, physical exam), collected as standard-of-care (SOC), included in their study chart. Participants will be started on sildenafil at V1. If tolerated, subjects will be maintained on sildenafil pre and post-LVAD implementation. On day 14 (+/- 2 days) subjects will have a RHC to evaluate right heart function post-LVAD implantation. Subjects will return to the VAD (Ventricular Assist Device) Clinic for regular visits following discharge until day 55 (EOS) for similar data collection. Subjects will keep a daily sildenafil dosage diary from hospital discharge until day 55. Subjects will receive a brief telephone call at day 85 post LVAD implantation to evaluate safety and outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years who are to receive durable (HeartMate II or III, or HeartWare HVAD) LVAD implantation for end-stage HF. Patients with all etiologies of HF will be included.
* Patients identified as having an increased risk for post-operative RHF using pre-operative hemodynamic assessment criteria, defined as the presence of ≥ 1 of the following: i) Central venous pressure (CVP):mean pulmonary capillary wedge pressure (PCWP) ratio ≥ 0.63 ii) RV stroke work index < 300 mmHg/mL/m2 iii) CVP ≥15 mmHg (CVP must be >8 mmHg if applying one of the other criteria) iv) Pre-operative PVR ≥ 3 Wood Units (240 dynes/cm5/sec)
* Systolic blood pressure ≥ 85 mmHg at study initiation
* Women of childbearing potential must have a negative pregnancy test. Women must not be breast feeding. Heterosexually active women of child bearing potential must use an effective method of contraception during the study.
* Ability to sign informed consent to participate

Exclusion Criteria:

* Preoperative INTERMACS level I or II
* Preoperative systemic hypotension with mean arterial pressure < 60 mmHg
* Planned insertion of RV support device (either temporary or permanent)
* Complex congenital heart disease where PVR measurement is not feasible or reliable (repaired or unrepaired)
* Right sided fixed or dynamic obstruction to blood flow (i.e., pulmonary stenosis) with resting gradient ≥ 10 mmHg.
* Previous organ transplantation
* Preoperative use of any oral pulmonary vasodilator therapy or oral/inhaled/nitrate therapy
* Patients requiring pre-operative hem - or peritoneal dialysis
* Pre-enrollment treatment with other pulmonary dilating agents such as other PDE5 inhibitors, endothelin antagonists, prostacyclin analogues. Use of postoperative nitric oxide will be permitted (although not concomitantly with the study medication) as clinically indicated in the postoperative setting
* Lack of ability to invasively measure right-sided pulmonary pressures
* Refusal or inability to sign informed consent
* Inability to accept preoperative study drug, or known sensitivity or allergy to sildenafil or any of its ingredients, or any other contra-indication to sildenafil as identified by product monograph
* Participation in any other current interventional (drug or device) study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance (PVR) | From baseline to postoperative day 14
  Change in PVR reported in Wood Units as measured invasively via right heart catheterization (RHC)

SECONDARY OUTCOMES:
Right heart failure (RHF) | From baseline to day 55 (end of study)
  Proportion of participants experiencing RHF defined as INTERMACS criteria: i) Requirement of continuous-flow right ventricular assist device (RVAD) implantation for hemodynamic support any time prior to study end
RHF | Postoperative day 14 to postoperative day 55 (end of study)
  Proportion of participants experiencing RHF defined as INTERMACS criteria: ii) Prolonged inotropic support beyond postoperative day 14 directed for clinical RHF
RHF | From baseline to postoperative day 55 (end of study)
  Proportion of participants experiencing RHF defined as INTERMACS criteria: iii) Discontinuation of study drug for the purpose of introduction of additional pulmonary vasodilator for the purpose of treatment of clinical RHF at any time during the study protocol
Inotrope requirement | From baseline to day 55 (study end)
  Proportion of patients requiring any inotrope medication at study end
ICU | From baseline to day 55 (end of study)
  Total number of hours in ICU by study end
Hospitalization | From baseline to day 55 (end of study)
  Total hospital length of stay by study end

OTHER OUTCOMES:
Safety: Drug interruptions | From baseline to day 55 (study end)
  Proportion of patients with temporary or permanent study drug interruptions
Safety: Renal | From baseline to day 55 (study end)
  Proportion of patients requiring renal replacement therapy or doubling of serum creatinine
Safety: All-cause mortality | From enrollment to day 85 (final SAE review)
  All-cause mortality at study end
Safety: Transfusion | From baseline to hospital discharge
  Total number of units of packed red cells transfused during hospital stay
Safety: GFR | From baseline fo day 55 (study end)
  Greatest percentage increase in glomerular filtration rate from baseline at any time during study
Safety: Mean arterial pressure | At ICU discharge and at day 55 (study end)
  Mean arterial pressure
Safety: Symptomatic hypotension | From baseline to day 55 (study end)
  Proportion of patients with > or = 1 episodes of symptomatic hypotension (syncope or orthostatic hypotension)
Safety: Liver enzymes | From baseline to day 55 (study end)
  Increase in hepatic enzymes > or = 2x baseline (preoperative) levels
Safety: Pump time | LVAD implantation day
  Total cardiac surgical bypass pump time
Safety: Adverse drug reactions | From baseline to day 85 (final SAE review)
  Any and all adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Howlett, FRCPC, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - St. Boniface Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fine NM, Litwin O, Kent WDT, Holloway DD, Roy J, Miller RJH, Chih S, Davey RA, Isaac DL, Sharma N, Lyons KJ, Howlett JG. Feasibility of Sildenafil for the Prevention of Right Heart Failure After Continuous-Flow Left Ventricular Assist Device Implantation: The REVAD Trial. Can J Cardiol. 2024 Apr;40(4):659-661. doi: 10.1016/j.cjca.2023.11.017. Epub 2023 Nov 22. No abstract available. PMID 37995907